CLINICAL TRIAL: NCT03839446
Title: Combination of Mitoxantrone, Etoposide and Gemtuzumab Ozogamicin (MEGO) for Patients With Acute Myeloid Leukemia Refractory to Initial Standard Induction Therapy
Brief Title: Phase II Study of the Combination of Mitoxantrone, Etoposide and Gemtuzumab Ozogamicin (MEGO) for Patients With Acute Myeloid Leukemia Refractory to Initial Standard Induction Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Redner, MD (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Robert Redner, MD, Professor of Medicine - Hematology/Oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 18-111
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: cytogenetic status; mitoxantrone; etoposide; gemtuzumab ozogamicin; bone marrow
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Mitoxantrone; Etoposide; Gemtuzumab

STUDY DESIGN:
Intervention Model Description: Open label single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mitoxantrone + etoposide + gemtuzumab ozogamicin (Experimental): 10 mg/m2 mitoxantrone days 1-5 + 100mg/m2 etoposide days 1-5 + 3mg/m2 gemtuzumab ozogamicin on day 6
  Interventions: Drug: mitoxantrone + etoposide + gemtuzumab ozogamicin

INTERVENTIONS:
Drug: mitoxantrone + etoposide + gemtuzumab ozogamicin — 10 mg/m2 mitoxantrone days 1-5 + 100mg/m2 etoposide days 1-5 + 3mg/m2 gemtuzumab ozogamicin on day 6.

SUMMARY:
This study is an open-label, single arm phase II study which will examine the efficacy and toxicity of the combination therapy of GO, mitoxantrone and etoposide in patients who did not respond to first line induction therapy.

DETAILED DESCRIPTION:
Eligible patients will be treated inpatient. Patients will receive mitoxantrone 10mg/m2 administered intravenous piggyback (IVPB) in 50ml 0.9% normal saline over 15 minutes on days 1-5 and etoposide 100 mg/m2 administered intravenously in 500 ml of 0.9% sodium chloride over 2 hours on days 1-5.

On day 6, patients will receive a single dose of GO 3mg/m2 (maximum dose 4.5mg). Patients will be pre-medicated 1 hour prior to the GO infusion with diphenhydramine 50mg administered orally or intravenously, acetaminophen 650 mg administered orally or intravenously and 1mg/kg methylprednisolone or an equivalent dose of alternative corticosteroid administered IV within 30 minutes prior to infusion of GO. GO will be administered intravenously in 50 ml (or other suitable volume resulting in a final GO concentration between 0.075 mg/mL to 0.234 mg/mL) of 0.9% sodium chloride over 2 hours. Doses of GO will be based on BSA calculated using actual body weight with a cap of 4.5mg. Vital signs will be recorded within one hour prior to the infusion and then every 30 minutes during the infusion and 30 minutes and one hour after completion of infusion. An additional dose of methylprednisolone 1 mg/kg IV may be given for any sign of infusion reaction, such as fever, chills, hypotension, or dyspnea occurring during the GO infusion or within 4 hours after the GO infusion.

For dose modifications based on kidney and liver function please see the treatment schema at the end of the study.

Supportive care including blood product transfusions, antiemetic medications, antiviral and antifungal medications, growth factor support, tumor lysis syndrome prophylaxis, or empiric antibiotics may be used at the clinical discretion of the provider.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and have the ability to provide written consent.
2. Age: ≥18 and ≤75 years-old
3. Patients with newly diagnosed AML based on the World Health Organization classification who have persistent disease after their first course treatment with an anthracycline and cytarabine (the diagnosis of persistent disease, which is defined as ≥10% blasts by morphology for this trial or >5% blasts if they have had an increase in blasts from the last bone marrow biopsy, will be based on their assessment after bone marrow aspiration and/or biopsy after initial treatment).
4. Patients with myelodysplastic syndrome (MDS) based on the World Health Organization classification who have persistent disease after their treatment with an anthracycline and cytarabine (the diagnosis of persistent disease, which is defined as ≥10% blasts by morphology for this trial or >5% blasts if they have had an increase in blasts from the last bone marrow biopsy, will be based on their assessment after bone marrow aspiration and/or biopsy after initial treatment).
5. CD33 expression in ≥ 30% of leukemic blasts on the bone marrow.
6. Eastern Cooperative Oncology Group Performance Status of 0 -2 (see Appendix I).
7. Patients must have the following laboratory values prior to beginning protocol treatment:

   * Calculated creatinine clearance ≥ 30 mL/min (using the Cockcroft-Gault equation CL creatinine = ((140-age) x body mass X 0.85 if female)/72 x creatinine where age is given in years, body mass is given in Kg and creatinine is given in mg/dl).
   * Aspartate aminotransferase (AST) ≤ 2.5 x upper normal limit.
   * Alanine aminotransferase (ALT) ≤ 2.5 x upper normal limit.
   * Total bilirubin ≤ 2 x upper normal limit. Note: As many eligible patients will be pancytopenic secondary to their disease or prior treatments, hematologic abnormalities will not be used as criteria for entry or exclusion.
8. Left ventricular ejection fraction (LVEF) ≥50 %.
9. Females of child-bearing potential must have a negative pregnancy test during screening and all subjects must agree to use an effective method of contraception. A woman is eligible to enter and participate in the study if she is of:

   1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who has had a hysterectomy or has had a bilateral oophorectomy (ovariectomy).
   2. Childbearing potential, has a negative serum pregnancy test during the screening period and agrees to avoid sexual activity or use contraception from screening through follow-up (method of birth control if the patient is not neutropenic include the use of a diaphragm, intrauterine device, contraceptive sponge and/or usage of male condom with a spermicide from the partner). A man with a female partner of childbearing potential is eligible to enter and participate in the study if he has either had a prior vasectomy or agrees to avoid sexual activity or use adequate contraception (as described above) from screening through follow-up.

Exclusion Criteria:

1. Patients with a diagnosis of Acute Promyelocytic Leukemia (APL) as defined by the World Health Organization.
2. Relapsed acute leukemia.
3. Bi-lineage or bi-phenotypic leukemia.
4. Prior use of mitoxantrone or etoposide or GO.
5. Previous allogeneic hematopoietic cell transplantation.
6. First induction course of acute myeloid leukemia with CPX-351.
7. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of treating investigator.
8. Has known history of active Hepatitis B (HBsAg reactive) or Hepatitis C (detectable HCV RNA).
9. Uncontrolled, life-threatening infection that is not responding to antimicrobial therapy.
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Patient may have not received any other investigational anti-neoplastic agents within 4 weeks from the start of therapy.
12. Concurrent active malignancy; exceptions include patients who have been disease free for 5 years, patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma, or patients with another malignancy with better prognosis than AML.
13. Women who are pregnant or breastfeeding.
14. Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory or cardiac disease).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2024-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Redner Robert, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All trial participants
Arm/Group | Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 59 [26.0 to 72.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Status [Count of Participants; unit: Participants] — Scoring:
  0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities; Up and about more than 50% of waking hours
  3. - Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. - Completely disabled; Cannot carry out any selfcare; Totally confined to bed or chair
  5. - Death
  Participants
    ECOG = 0 | 1
    ECOG = 1 | 15
Cytogenetic Status [Count of Participants; unit: Participants] — Number of patients with Poor, Intermediate, or Favorable chromosomal status (potential predictor of outcome).
  Participants
    Poor | 13
    Intermediate / Favorable | 3
Percent bone marrow blasts [Median (Full Range); unit: Percent bone marrow blasts] — Percent of blasts present in the bone marrow.
  Percent bone marrow blasts | 50.9 [8.00 to 89.0]
Percent CD33 expression in leukemia blasts [Median (Full Range); unit: % CD33 expression] — Percentage of CD33 expression in leukemia blasts.
  % CD33 expression | 100 [36.0 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate
Description: The estimated percentage of patients with Complete Responses (CR / total response-evaluable patients x 100). CR in AML is defined as: 1. Normal values for absolute neutrophil count (>1000/microL), platelet count (>100,000/microL), independence from red cell transfusion. 2. Bone marrow biopsy reveals no clusters or collections of blast cells. Extramedullary leukemia (eg, central nervous system or soft tissue involvement) must be absent. 3. Bone marrow aspiration reveals normal maturation of all cellular components (ie, erythrocytic, granulocytic, and megakaryocytic series). No requirement for bone marrow cellularity. 4. < 5 percent blast cells are present in the bone marrow, and none can have a leukemic phenotype (eg, Auer rods). 5. The absence of a previously detected clonal cytogenetic abnormality (ie, complete cytogenetic remission, CRc) confirms the morphologic diagnosis of CR but is not currently required.
Time Frame: Up to six weeks
Population: To be evaluable for clinical response, a patient must have received a total of 5 days of mitoxantrone and etoposide, received 1 dose of GO and had a follow-up bone marrow biopsy to evaluate the response to therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin
Number analyzed (Participants) | 14
percentage of participants | 36 [15 to 100]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: The length of time during and after the treatment that a patient lives with Acute Myeloid Leukemia disease that does not progress.
Time Frame: Up to five years
Population: Patients who were evaluable for response to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin
Number analyzed (Participants) | 16
months | 3.27 [0.92 to 39.43]
Statistical Analysis 1: Comparison: Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin; Cytogenetic status; Test type: Superiority; p = 0.777, Regression, Cox; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.18 to 3.65] — Intermediate / Favorable vs Poor
Statistical Analysis 2: Comparison: Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin; Percent of blasts present in the bone marrow; Test type: Superiority; p = 0.200, Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.96 to 1.01]
Statistical Analysis 3: Comparison: Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin; % CD33 expression in leukemia blasts; Test type: Superiority; p = 0.014, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.94 to 0.99]

3. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the start of treatment that patients are still alive.
Time Frame: Up to five years
Population: All treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin
Number analyzed (Participants) | 16
months | 17.4 [7.23 to NA] — Upper bound of the 95% CI was not reached due to low number of events.
Statistical Analysis 1: Comparison: Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin; Cytogenetic status; Test type: Superiority; p = 0.801, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.17 to 3.86] — Intermediate / Favorable vs Poor
Statistical Analysis 2: Comparison: Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin; % bone marrow blasts; Test type: Superiority; p = 0.168, Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.95 to 1.01]
Statistical Analysis 3: Comparison: Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin; % CD33 expression in leukemia blasts; Test type: Superiority; p = 0.015, Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.94 to 0.99]

ADVERSE EVENTS:
Time Frame: Adverse Events monitored for 4 weeks after discharge and then every 2 weeks until count recovery (defined as ANC ≥ 1000 with or without PLT ≥ 100,000), up to 4 years. All-Cause Mortality monitored up to 4 years.
Arm/Group | Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin
All-Cause Mortality (participants affected / at risk) | 7/16
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin (N=16)
Sepsis (Blood and lymphatic system disorders) | 1 (16)
Platelet count decreased (Investigations) | 1 (16)
Nervous system disorders - Other, specifyEpidural, subdural, subarachnoid hematoma (Nervous system disorders) | 1 (16)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitoxantrone + Etoposide + Gemtuzumab Ozogamicin (N=16)
Anemia (Blood and lymphatic system disorders) | 16
Blood and lymphatic system disorders - Other, specifyDecreased WBC (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specifyIncreased AST (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specifyIntermittent Decreased Platelets (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specifyLow ACL (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specifyLow ANC (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 13
Cardiac arrest (Cardiac disorders) | 1
Cardiac disorders - Other, specifyPVC/SVT (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 4
Ventricular fibrillation (Cardiac disorders) | 1
Dry eye (Eye disorders) | 1
Eye disorders - Other, specifyL eye hemorrhage (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specifyHemorrhoidal Pain (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specifyMelena (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 9
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 5
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 7
General disorders and administration site conditions - Other, specifydry lips (General disorders) | 1
Generalized edema (General disorders) | 3
Hypothermia (General disorders) | 1
Localized edema (General disorders) | 1
Malaise (General disorders) | 2
Multi-organ failure (General disorders) | 2
Pain (General disorders) | 6
Hepatic failure (Hepatobiliary disorders) | 1
Immune system disorders - Other, specifymyalgia (Immune system disorders) | 1
Bacteremia (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 2
Infections and infestations - Other, specifyPalmar plantar erythrodysesthesia (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Thrush (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specifyacute kidney injury (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Fibrinogen decreased (Investigations) | 4
INR increased (Investigations) | 6
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 12
Weight gain (Investigations) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 5
Acidosis (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hyperphosphatemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Nervous system disorders - Other, specifyBradycardia (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 4
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifydry nose (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyR Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specifyShortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 3
Phlebitis (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT03839446/Prot_SAP_000.pdf